CLINICAL TRIAL: NCT02157350
Title: A Prospective Study to Identify Predictive Factors for Progression and Regression of Proliferative Diabetic Retinopathy in Patients Receiving Standard Panretinal Laser Photocoagulation.
Brief Title: The Individually Marked Panretinal lasEr phoTokoagUlation for Proliferative Diabetic Retinopathy Study - DETECT
Acronym: IMPETUS-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); National University of Singapore (Other); Yamagata University (Other)
Responsible Party: Principal Investigator, Thomas Lee Torp, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUH-4202-ID-2018; S-20140046 (Other: The Danish National Committee on Health Research Ethics)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Eye Diseases; Proliferative Diabetic Retinopathy; Retinal Vessel Geometry; Retinal Oxymetry; Retina Ischemia; Panretinal Photocoagulation; Lasers, Semiconductor; Fluorescein Angiography
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Intervention Model Description: Panretinal photocoagulation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panretinal Laser Photocoagulation (Experimental): See interventional description.
  Interventions: Procedure: Panretinal laser photocoagulation

INTERVENTIONS:
Procedure: Panretinal laser photocoagulation — Panretinal photocoagulation. Laser energy is given to the retina in two sittings, carefully avoiding the macular. The energy are placed 2 to 3 disc diameters away from the macula and the disc outside the arcades and extended peripherally upto the equator and beyond.
  Other Names: NAVILAS laser; Retinal Laser Photocoagulation

SUMMARY:
The purpose of this study is to determine the threshold level of proliferative diabetic retinopathy progression and regression after standard panretinal photocoagulation. Predictors of progression and regression will be identified which will include retinal vessel geometry (caliber, fractals and tortuosity), retinal vessel oxygen saturation and retinal areas of non-perfusion.

DETAILED DESCRIPTION:
IMPETUS 2018 - DETECT is a six-month prospective study involving 90 treatment-naïve diabetes patients with proliferative diabetic retinopathy (PDR) referred for panretinal laser photocoagulation (PRP) treatment to the Department of Ophthalmology, Odense University Hospital between July 1st 2014 and June 30th 2015.

Project information will be given prior to the study to the ophthalmological departments of and to all private practicing ophthalmologists in the Region of Southern Denmark. Patients will at baseline have a standard examination that will include wide-field fundus photography, wide-field fluorescein angiography and spectral domain optical coherence tomography (SD-OCT) in order to confirm the diagnosis of PDR. If they meet the criteria of inclusion and not those of exclusion, they will be informed of the study verbally and writing and offered the chance to participate. Prior to the first session of PRP patients enrolled in the study will receive the rest of the baseline examinations including retinal oximetry. Standard PRP treatment will be given in two sessions by a trained doctor.

Patients will be re-examined at month 3 and 6 and progression/regression of PDR will be evaluated by measuring the amount of fluorescein leakage by wide-field fluorescein angiography at 1, 5 and 10 minutes. For patients with regression, supplementary PRP will be offered. After the final examination at month 6, patients will be referred back to their primary ophthalmologist.

A study nurse and a photographer will be assigned to the project. All examinations will be standardized and the study crew will be fully certified. Data will be analyzed with respect to the endpoint of the study (Stata 13, StataCorp, College Station, Texas) and also used to create the algorithm to be used for individualized treatment in IMPETUS 2018 - TREAT.

In the Region of Southern Denmark it is estimated that 200 treatment naïve patients with PDR will be referred for treatment annually. With an estimated participation rate of 50% and a subsequent dropout rate of 10%, IMPETUS 2018 - DETECT will include 90 patients. A traditional power calculation is not feasibly due to the design of the study with multiple outcomes studies.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Proliferative diabetic retinopathy of one or both eyes

Exclusion Criteria:

* Diabetic macular edema on current eye
* Earlier PRP treatment on current eye
* Cataract demanding treatment on current eye
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Proliferative diabetic retinopathy progression/regression. | Change from baseline in proliferative diabetic retinopathy at 6 months
  Progression/regression of proliferative diabetic retinopathy will be evaluated by measuring the amount of fluorescein leakage by wide-field fluorescein angiography at 1, 5 and 10 minutes. These measurements will be performed at baseline, and during followup after panretinal photocoagulation (3 months and 6 months).

SECONDARY OUTCOMES:
Retinal vessel geometry (caliber, fractals and tortuosity) | Measurements assessed at baseline and 3 and 6 months after panretinal laser photocoagulation.
  Change in vessel geometry:
  Caliber: Using a computerised program - SIVA / IVAN. Fractals: Using a computerised program - SIVA. Tortuosity: Using a computerised program - SIVA

OTHER OUTCOMES:
Retinal vessel oxygen saturation | Measurements assessed at baseline and 3 and 6 months after panretinal laser photocoagulation.
  Oxymap T1 with the Oxymap Analyser. Non-invasively measuring the vessel saturation of both arterioles and venules in percentage.
Retinal areas of non-perfusion. | Measurements assessed at baseline and 3 and 6 months after panretinal laser photocoagulation.
  Using wide-field fluorescein angiography

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Torp, MD, Principal Investigator — Research Unit of Ophthalmology, University of Southern Denmark; Joakob Grauslund, DMSci, PhD, Study Director — Research Unit of Ophthalmology, University of Southern Denmark; Tundo Peto, PhD,FHCO, Study Chair — NIHR Biomedical Research Centre at Moorfields Eye Hospital NHS; Tien Y Wong, PhD, Study Chair — Department of Ophthalmology National University of Singapore; Ryo Kawasaki, PhD, Study Chair — Department of Public Health Ophthalmology, Yamagata
Locations (1):
- Research Unit of Ophthalmology, Clinical Institute, University of Southern Denmark, Department of Ophthalmology, Odense University Hospital., Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grauslund J, Green A, Sjolie AK. Blindness in a 25-year follow-up of a population-based cohort of Danish type 1 diabetic patients. Ophthalmology. 2009 Nov;116(11):2170-4. doi: 10.1016/j.ophtha.2009.04.043. Epub 2009 Sep 10. PMID 19744716
- [Background] Grauslund J, Green A, Sjolie AK. Prevalence and 25 year incidence of proliferative retinopathy among Danish type 1 diabetic patients. Diabetologia. 2009 Sep;52(9):1829-35. doi: 10.1007/s00125-009-1450-4. Epub 2009 Jul 12. PMID 19593541
- [Background] Stefansson E. Ocular oxygenation and the treatment of diabetic retinopathy. Surv Ophthalmol. 2006 Jul-Aug;51(4):364-80. doi: 10.1016/j.survophthal.2006.04.005. PMID 16818083
- [Background] Preliminary report on effects of photocoagulation therapy. The Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1976 Apr;81(4):383-96. doi: 10.1016/0002-9394(76)90292-0. PMID 944535
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Ferris FL 3rd, Podgor MJ, Davis MD. Macular edema in Diabetic Retinopathy Study patients. Diabetic Retinopathy Study Report Number 12. Ophthalmology. 1987 Jul;94(7):754-60. doi: 10.1016/s0161-6420(87)33526-2. PMID 3658347
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Klein R, Klein BE, Moss SE, Wong TY, Hubbard L, Cruickshanks KJ, Palta M. The relation of retinal vessel caliber to the incidence and progression of diabetic retinopathy: XIX: the Wisconsin Epidemiologic Study of Diabetic Retinopathy. Arch Ophthalmol. 2004 Jan;122(1):76-83. doi: 10.1001/archopht.122.1.76. PMID 14718299
- [Background] Rogers SL, Tikellis G, Cheung N, Tapp R, Shaw J, Zimmet PZ, Mitchell P, Wang JJ, Wong TY. Retinal arteriolar caliber predicts incident retinopathy: the Australian Diabetes, Obesity and Lifestyle (AusDiab) study. Diabetes Care. 2008 Apr;31(4):761-3. doi: 10.2337/dc07-1622. Epub 2008 Jan 9. PMID 18184895
- [Background] Klein R, Klein BE, Moss SE, Wong TY. Retinal vessel caliber and microvascular and macrovascular disease in type 2 diabetes: XXI: the Wisconsin Epidemiologic Study of Diabetic Retinopathy. Ophthalmology. 2007 Oct;114(10):1884-92. doi: 10.1016/j.ophtha.2007.02.023. Epub 2007 May 30. PMID 17540447
- [Background] Grauslund J, Hodgson L, Kawasaki R, Green A, Sjolie AK, Wong TY. Retinal vessel calibre and micro- and macrovascular complications in type 1 diabetes. Diabetologia. 2009 Oct;52(10):2213-7. doi: 10.1007/s00125-009-1459-8. Epub 2009 Jul 18. PMID 19618163
- [Background] Grauslund J, Green A, Kawasaki R, Hodgson L, Sjolie AK, Wong TY. Retinal vascular fractals and microvascular and macrovascular complications in type 1 diabetes. Ophthalmology. 2010 Jul;117(7):1400-5. doi: 10.1016/j.ophtha.2009.10.047. Epub 2010 Feb 21. PMID 20176399
- [Background] Sasongko MB, Wong TY, Nguyen TT, Cheung CY, Shaw JE, Wang JJ. Retinal vascular tortuosity in persons with diabetes and diabetic retinopathy. Diabetologia. 2011 Sep;54(9):2409-16. doi: 10.1007/s00125-011-2200-y. Epub 2011 May 29. PMID 21625945
- [Background] Jorgensen CM, Hardarson SH, Bek T. The oxygen saturation in retinal vessels from diabetic patients depends on the severity and type of vision-threatening retinopathy. Acta Ophthalmol. 2014 Feb;92(1):34-9. doi: 10.1111/aos.12283. Epub 2013 Dec 16. PMID 24330421
- [Background] Ober MD, Kernt M, Cortes MA, Kozak I. Time required for navigated macular laser photocoagulation treatment with the Navilas. Graefes Arch Clin Exp Ophthalmol. 2013 Apr;251(4):1049-53. doi: 10.1007/s00417-012-2119-0. Epub 2012 Aug 7. PMID 22868445
- [Background] Kernt M, Cheuteu R, Vounotrypidis E, Haritoglou C, Kampik A, Ulbig MW, Neubauer AS. Focal and panretinal photocoagulation with a navigated laser (NAVILAS(R)). Acta Ophthalmol. 2011 Dec;89(8):e662-4. doi: 10.1111/j.1755-3768.2010.02017.x. Epub 2010 Oct 14. No abstract available. PMID 20946326
- [Background] Hardarson SH. Retinal oximetry. Acta Ophthalmol. 2013 Aug;91(5):489-90. doi: 10.1111/aos.12239. No abstract available. PMID 23844858
- [Background] Geirsdottir A, Palsson O, Hardarson SH, Olafsdottir OB, Kristjansdottir JV, Stefansson E. Retinal vessel oxygen saturation in healthy individuals. Invest Ophthalmol Vis Sci. 2012 Aug 13;53(9):5433-42. doi: 10.1167/iovs.12-9912. PMID 22786895
- See also: The Regional Scientific Ethical Committees for Southern Denmark — http://komite.regionsyddanmark.dk/wm258128
- See also: The Danish Data Protection Agency — http://www.datatilsynet.dk/
- See also: University of Southern denmark — http://www.sdu.dk/en/forskning/phd